CLINICAL TRIAL: NCT03849131
Title: Patient-Reported AutoImmunity Secondary to Cancer immunothErapy
Acronym: PRAISE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6994
Record Dates: First submitted 2019-01-09; First posted 2019-02-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Opportunistic Autoimmune Diseases
Keywords: monoclonal anti-PD-1 immunotherapy; monoclonal anti-CTLA-4 immunotherapy; checkpoint inhibitors; autoimmune manifestations; patient reported outcome; oncology
MeSH Terms: conditions — Neoplasms | interventions — Biological Specimen Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Biological collection — Blood samples will be collected only once at enrollment, before initiation of a checkpoint inhibitor.
  It will include:
  * DNA samples collection
  * RNA samples collection
  * Blood sample collection
  Other Names: Biobank

SUMMARY:
This is a real life observational longitudinal study aiming to identify autoimmune manifestations in patients treated with "checkpoint inhibitors" in mono or combo therapy in real life.

The study is based on patients reported experience validated by physician, recruited in cancer centers in France with another data collection from a French healthcare data claims database and a biological collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (over 18 year old) in France (DOM/TOM included), starting a monoclonal anti-PD-1 and/or anti-CTLA-4 immunotherapy for a cancer, whatever the cancer, within the Marketing Authorization.

  * As this research will be funded by BMS, for the e-Cohort, we will consider only patients treated by a BMS monoclonal antibody, to date: Ipilimumab (YERVOY©), Nivolumab (OPDIVO©) and Combo according to SmPCs.
  * All patients (anonymous) with a reimbursed checkpoint inhibitor drug in SNDS will be included for the healthcare database claims study.
* Included patients should be able to understand and fill in questionnaires in French and should give informed consent and contact details, they should be able to read and answer emails in French.

  * French Healthcare insurance beneficiary, whatever the scheme is.

Exclusion Criteria:

* Patients in all interventional clinical trials, with exclusion from other studies specifically mentioned
* Patients deprived of liberty or guardianship
* Women of childbearing potential with a desire of becoming pregnant
* Major patients under tutorship.
* Patients with dementia or drug addiction
* Patients with no regular access to internet and phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
incidence of severe autoimmune manifestations in patients treated with BMS checkpoint inhibitors. | 2 years after inclusion
  Severe autoimmune manifestations is defined by :
  * Discontinuation (temporary or definitive) of the cancer immunotherapy related to Autoimmunity
  * or requirement for treatment due to auto-immune manifestations according to expert judgement
  * or hospitalization for autoimmune manifestations
  * or death related to autoimmune manifestations

SECONDARY OUTCOMES:
Comparison of the age for the two groups of patients | 2 years after inclusion
  Comparison of the age for the two groups of patients (one who develop severe autoimmune manifestations, one who does not develop severe autoimmune manifestations)
Comparison of the gender for the two groups of patients | 2 years after inclusion
  Comparison of the gender for the two groups of patients (one who develop severe autoimmune manifestations, one who does not develop severe autoimmune manifestations)
Comparison of the body-mass index for the two groups of patients | 2 years after inclusion
  Comparison of the body-mass index for the two groups of patients (one who develop severe autoimmune manifestations, one who does not develop severe autoimmune manifestations)
Comparison of the types of cancer for the two groups of patients | 2 years after inclusion
  Comparison of the types of cancer for the two groups of patients (one who develop severe autoimmune manifestations, one who does not develop severe autoimmune manifestations)
Comparison of the number of previous lines of chemotherapy for the two groups of patients | 2 years after inclusion
  Comparison of the number of previous lines of chemotherapy for the two groups of patients (one who develop severe autoimmune manifestations, one who does not develop severe autoimmune manifestations)
Event-free survival of patients | 2 years after inclusion
  Time that passes before first appearance of Opportunistic Autoimmunity Secondary to cancer Immunotherapy. The baseline is the onset of cancer immunotherapy.
Description of flares or worsening of pre-existing autoimmune diseases | 2 years after inclusion
  Pre-existing autoimmune disease will be defined by expert judgement on history of autoimmunity ongoing activity and blood analysis (preexisting autoantibodies will be investigated using biobanked serum)
Comparison of baseline predictive factors of autoimmune manifestations for the two groups of patients | 2 years after inclusion
  Assessment of the prevalence of preexisting autoantibodies before immune checkpoint inhibitor initiation for the two groups of patients (one who develop severe autoimmune manifestations, one who does not develop severe autoimmune manifestations)
Changes in patients' quality of life over time and the impacts of OASI | 2 years after inclusion
  EQ-5D-5L general quality of life scores
Changes in patients' quality of life over time and the impacts of OASI | 2 years after inclusion
  EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques-Eric GOTTENBERG, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Hopitaux universitaires de strasbourg, Strasbourg, Alsace, France